CLINICAL TRIAL: NCT01064180
Title: Randomized,2-way Crossover, Bioequivalence Study of Carvedilol 25 mg Film-coated Tablets and COREG® 25 mg Film-coated Tablets Administered as 1 x 25 mg Film-coated Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Carvedilol 25 mg Film-coated Tablets, Bioequivalence Study of Dr. Reddys Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Assistanct Manager - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02118
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol Tablets 25 mg of Dr Reddys Laboratories Limited
  Interventions: Drug: Carvedilol
- Coreg (Active Comparator): Coreg Tablets 25 mg of GlaxoSmithKline
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol Tablets 25 mg
  Other Names: Coreg Tablets 25 mg

SUMMARY:
Carvedilol 25 mg Film-coated Tablets, Bioequivalence Study of Dr. Reddys Under Fed Conditions

DETAILED DESCRIPTION:
A Randomized,Two-way Crossover, Bioequivalence Study of Carvedilol 25 mg Film-coated Tablets and COREG® 25 mg Film-coated Tablets administered as 1 x 25 mg Film-coated Tablet in Healthy Subjects Under Fed Conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may be done using different media (e.g. radio, newspaper, Anapharm Inc. Website, Anapharm Inc. volunteers' data base). Subjects must meet all of the following criteria in order to be included in the study:

* Subjects will be females and/or males, smokers and non-smokers, 18 years of age & older.
* Female subjects will be post-menopausal/surgically sterilized.

  * Post-menopausal status is defined as absence of menses for the past 12 months or hysterectomy with bilateral oophorectomy at least 6 months ago.
  * Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses/surgery within 4 weeks prior to the administration of study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Subjects with a clinically significant history of second- or third-degree AV block, sick sinus syndrome or severe bradycardia or in patients with cardiogenic shock who have decompensated heart failure.
* Subjects with history of hepatic failure.
* Presence or history of liver disease, cardiovascular disease, diabetes, hyperthyroidism aDd peripheral vascular disease.
* Positive urine drug screen or positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure <ll0 or over 140 mmHg, or diastolic blood pressure <70 or over 90 mmHg; or heart rate <60 or over 100 bpm) at screening.
* Subjects with BMI ≥30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* History of allergic reactions to carvedilol or other beta-blocking agents (e.g. propranolol, labetalol, acebutolol, atenolol, esmolol, metoprolol, oxprenolol, timolol, pindolol, betaxolol, levobunolol and nadolol).
* History of pulmonary or bronchospastic disease (including asthma).
* Subjects with pheochromocytoma.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin,ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural products, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:
* less than 300 mL of whole blood within 30 days or
* 300 mL to 500 mL of whole blood within 45 days or
* more than 500 mL of whole blood within 56 days.
* Smoking more than 25 cigarettes per day.
* Subjects who have consumed food or beverages containing grapefruit (e.g. fresh, canned,or frozen) within 7 days prior to administration of the study medication.

Additional exclusion criteria for females only:

• Breast-feeding subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-05; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Carvedilol Tablets, 25 mg Bioequivalence Study Of Dr Reddys under non-fasting condition | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bircell, MD, Principal Investigator — Anapharm Inc, Canada, GIV 2K8; Benoit Girard, MD, Study Director — Anapharm Inc, Canada, H3X 2H9